CLINICAL TRIAL: NCT05255016
Title: Safety and Effectiveness of the PXL Platinum 330 System With Riboflavin Solution for Refractory Corneal Ulcers
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peschke GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PXL-330-02A
Record Dates: First submitted 2022-01-25; First posted 2022-02-24 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Keratitis; Corneal Ulcer
MeSH Terms: conditions — Keratitis; Corneal Ulcer | interventions — Riboflavin; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: Simple block randomization will be used to assign subjects in a 1:1 ratio to 2 treatment arms. Subjects will be randomized consecutively (not stratified by site) to ensure balance between the treatment arms at any point in the study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Standard of care + Sham CXL + Artificial Tears (Sham Comparator): Standard-of-care treatment and Sham CXL and administration of artificial tears.
  Interventions: Other: Sham CXL + Artificial Tears
- Standard of care + CXL + Riboflavin 0.25% TE Solution (Experimental): Standard of care treatment and the experimental combination product. The PXL Platinum 330 Illumination System is a portable electronic medical device. The device's light emitting diode (LED) is used to deliver a metered dose of UV-A light to a targeted treatment area for illuminating the cornea during corneal collagen CXL. The riboflavin solution is an isotonic (0.9%) sodium chloride solution containing 0.25% riboflavin, 1% hydroxypropylmethylcellulose, and 0.007% benzalkonium chloride, adjusted to a pH of 7.0, and packaged in 2 mL sterile syringes for topical ophthalmic use.
  Interventions: Combination Product: PXL Platinum 330 system + Riboflavin 0.25% TE Solution

INTERVENTIONS:
Combination Product: PXL Platinum 330 system + Riboflavin 0.25% TE Solution — Standard-of-care therapy (antifungal drops or fortified antibiotics and empiric antibiotic drops). In addition CXL + Riboflavin 0.25% TE solution.
  After topical anesthesia, the surgeon or trained designee will apply topical riboflavin (1 drop every 2 min for 40 min with PESCHKE TE solution [0.25%], or longer as needed to assure adequate corneal penetration). At the end of this pre-treatment period, the eye will be examined at the slit lamp with the blue filter for the presence of riboflavin throughout the stroma. When sufficient corneal riboflavin penetration is confirmed, the eye will be aligned under the PXL Platinum 330 light. The correct aperture setting (3 to 12 mm) will be selected for the size of the eye and area needing to be treated (2 mm larger than the maximal ulcer diameter), and the eye will be irradiated at 18 mW/cm2, with pulsed mode (5 seconds on, 5 seconds off) for 10 min, during which time instillation of riboflavin will continue (1 drop every 2 min).
  Arms: Standard of care + CXL + Riboflavin 0.25% TE Solution
Other: Sham CXL + Artificial Tears — Standard-of-care therapy (antifungal drops or fortified antibiotics and empiric antibiotic drops). In addition, for subjects in the sham group, artificial tears (1 drop every 2 min for 40 min) will be administered. after instillation of artificial tears, the eye will be aligned under the PXL Platinum 330 light. The instrument will be kept off and the subject will be kept under the device for 10 min during which time instillation of artificial tears will be performed (1 drop every 2 min) to maintain corneal hydration. The operator will keep track of sham exposure time independently to confirm the actual duration.
  Arms: Standard of care + Sham CXL + Artificial Tears

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of using the PXL Platinum 330 System with riboflavin solution for performing corneal collagen crosslinking (CXL) for the treatment of refractory corneal ulcers. The PXL Platinum 330 System is a combination product consisting of an ultraviolet-A (UV-A) 365 nm wavelength light source (PXL Platinum 330 Illumination System) and riboflavin (Peschke Riboflavin 0.25% Transepithelial Solution) administered in conjunction with the UV-A light as a photosensitizer.

The PXL Platinum 330 System is intended to induce corneal collagen CXL to improve the biomechanical properties of the cornea by strengthening the corneal tissue in the anterior stroma. Corneal collagen CXL is performed by pretreating the cornea with riboflavin 0.25% ophthalmic solution beginning 40 min before UV-A light exposure to saturate the corneal tissue with the riboflavin photosensitizer. The cornea is then irradiated with UV-A light (365 nm) at an irradiance of 18 mW/cm2 (5 seconds on, 5 seconds off) for 10 min. Exposure of the cornea to this UV-A light regimen after topical administration of riboflavin (0.25%) has been shown to induce CXL of the corneal collagen fibrils, with a resultant increase in tensile strength and diameter of the collagen fibrils. Clinically, CXL has been shown to stabilize the corneal curvature in eyes with progressive keratoconus, with no significant change in the refractive index of the cornea. Numerous reports and a few clinical trials have also shown benefit in aiding resolution of infective corneal ulcers.

DETAILED DESCRIPTION:
This is a prospective, 2-arm parallel-group, single-blind, randomized multicenter study to determine the safety and effectiveness of the PXL Platinum 330 System for performing CXL in eyes with refractory corneal ulcers. Subjects with a history of non-resolving infective corneal ulcers will be evaluated initially for suitability as a candidate for CXL. Subjects who are candidates for CXL will be asked to participate in this study and will undergo the required screening procedures to determine study eligibility. Informed consent will be obtained from each subject before performance of any required study procedures that are not part of the investigator's routine examination. After completing screening procedures, the diagnosis for each eligible eye will be confirmed. Subjects will be randomized to 1 of 2 groups:

1. Group 1: Standard-of-care therapy (anti fungal drops if there is clinical suspicion for fungus, fortified antibiotics if corneal culture is positive for a specific organism sensitive to a fortified antibiotic, and empiric antibiotic drops based on community prevalence if corneal culture is negative and there is no clinical suspicion for fungus)
2. Group 2: Standard-of-care therapy + CXL

Eyes undergoing CXL will have topical anesthetic administered and then have topical riboflavin instilled onto the cornea every 2 min (or longer as needed to assure adequate corneal penetration), after which the cornea will be exposed to UV-A pulsed light 18 mW/cm2 for 10 min. Riboflavin instillation will continue every 2 min during CXL. The CXL procedures will be performed on an outpatient basis using the PXL Platinum 330 System (UV-A light source and riboflavin solution). All use of the PXL Platinum 330 System will be in accordance with this protocol and the general instructions provided by the manufacturer (PESCHKE) in the PXL Platinum 330 Illumination System Operator's Manual. All subjects will be evaluated at Screening/Baseline, Day 0 (Randomization/Treatment), Day 1, Day 3 ( +/- 1 day), Week 1 ( +/- 2 days), Week 2 ( +/- 2 days), Week 4 ( +/- 3 days), and Week 6 ( +/- 4 days) after treatment. Efficacy monitoring throughout the study will include observations at appropriate times for re-epithelialization, size of infection, and corneal culture results. Safety monitoring throughout the study will include observations at appropriate times for pain, IOP, BSCVA, corneal scar size, AEs, clinically significant findings on ophthalmic examination, dilated fundus examination, and slit lamp examination. After treatment, subjects will be followed at the treating physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Central corneal ulcer or hypopyon, and/or failure to improve within 24 hours of initiating conventional antibiotic eyedrops (eg, quinolone, polymyxin/trimethoprim, erythromycin, or other non-fortified antibiotics) or failure to completely re-epithelialisation within 1 week of initiating conventional antibiotic drops
3. Consent to a corneal culture for bacterial keratitis (suspected keratitis is defined as a corneal epithelial defect of any size with an infiltration of the underlying stroma)
4. Signed written informed consent
5. Willingness and ability to comply with schedule for follow-up visits
6. Minimum corneal thickness >300 μm

Exclusion Criteria:

1. Presence of a perforated corneal ulcer
2. Presence of a corneal ulcer that has produced a descemetocele
3. Presence of a corneal ulcer deeper than 50% depth or 275 μm in the cornea
4. Any active ocular infection other than the central corneal ulcer or hypopyon to be treated
5. Suspicion of amoebic or viral keratitis requiring treatment with topical anti- amoebic or topical antiviral ophthalmic medications
6. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye(s) for future complications. This may include history of or active corneal disease (eg, herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, acanthamoeba, etc.)
7. Uncontrolled systemic disease, especially a collagen-vascular or rheumatologic condition that could contribute to the corneal condition
8. Pregnancy (or plan to become pregnant) or lactation during the course of the study
9. A known sensitivity to study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-11-24 (Estimated); Study Completion 2024-02-24 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the safety and effectiveness of corneal collagen CXL (performed using the PXL-Platinum 330 system with riboflavin solution) for treating refractory corneal ulcers. | Week 2 (#+/- 2 study days).
  Primary Outcome Measure:
  1. The composite primary endpoint outcome would be the proportion of patients in the treated group, compared to the control group, who achieve all three of the following components:
     * complete re-epithelialization at week 2, defined as absence of corneal fluorescein staining noted with the blue light of the slit lamp by the investigator.
     * no expansion of infiltrate from baseline to week 2. The size of the infiltrate will be reviewed by the investigator using the slit lamp exam and compared to baseline measures to assess expansion of the infiltrate.
     * a negative corneal culture at week 2
  2. Each of the components of this composite endpoints is a binary outcome (yes or no), and are NOT measured as units of measure.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Viscuso, Study Director — Peschke GmbH; Bala Ambati, Principal Investigator — Pacific Clear Vision Institute
Locations (12):
- United States (12):
  - Colorado Eye Consultants, Littleton, Colorado
  - Gorovoy M.D Eye Specialists, Fort Myers, Florida
  - Bay Area Eye Institute, Tampa, Florida
  - Price Vision Group, Indianapolis, Indiana
  - The cornea & Laser Eye Institute-NJ, Teaneck, New Jersey
  - SightMD, Babylon, New York
  - Prisma Health Opthalmology, Columbia, South Carolina
  - Woolfson Eye, Chattanooga, Tennessee
  - Houston Eye Associates, Houston, Texas
  - San Antonio Eye Center, Lackland Air Force Base, Texas
  - Milwaukee Eye Surgeons, Milwaukee, Wisconsin
  - Valley Eye, Oshkosh, Wisconsin

IPD SHARING:
Plan to Share IPD: No